CLINICAL TRIAL: NCT03197857
Title: Determination of Factors Influencing the Physical Condition of Obese Patients Following Bariatric Surgery. Randomized Controlled Trial
Brief Title: Physical Condition and Bariatric Surgery
Acronym: CaPaCITy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CHU-320; 2016-A01432-49 (Other: 2016-A01432-49)
Record Dates: First submitted 2017-05-04; First posted 2017-06-23 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Obese Patients With Bariatric Surgery
Keywords: Bariatric surgery; Morbid obesity; Physical condition; Muscle; 6-minute walking test; Protein supplementation; Physical activity program
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Masking Description: open
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Control (Experimental): Physical condition will be evaluated in obese patients before surgery and 1, 4, 6, 12, 18 and 24 months after surgery.
  Between 1 and 4 months after surgery, participants will be assigned to one of the postoperative care groups:
  * Control
  * Control + protein supplementation
  * Training in aquabike
  * Training in aquabike + protein supplementation
  * Bicycle training
  * Bicycle training + protein supplementation
  Interventions: Behavioral: Physical activity program : without protein supplementation
- Control + protein supplementation (Experimental): Physical condition will be evaluated in obese patients before surgery and 1, 4, 6, 12, 18 and 24 months after surgery.
  Between 1 and 4 months after surgery, participants will be assigned to one of the postoperative care groups:
  * Control
  * Control + protein supplementation
  * Training in aquabike
  * Training in aquabike + protein supplementation
  * Bicycle training
  * Bicycle training + protein supplementation
  Interventions: Behavioral: Physical activity program : with protein supplementation
- Training in aquabike (Experimental): Physical condition will be evaluated in obese patients before surgery and 1, 4, 6, 12, 18 and 24 months after surgery.
  Between 1 and 4 months after surgery, participants will be assigned to one of the postoperative care groups:
  * Control
  * Control + protein supplementation
  * Training in aquabike
  * Training in aquabike + protein supplementation
  * Bicycle training
  * Bicycle training + protein supplementation
  Interventions: Behavioral: Physical activity program : aquabike; Behavioral: Physical activity program : without protein supplementation
- - Training in aquabike + protein supplementation (Experimental): Physical condition will be evaluated in obese patients before surgery and 1, 4, 6, 12, 18 and 24 months after surgery.
  Between 1 and 4 months after surgery, participants will be assigned to one of the postoperative care groups:
  * Control
  * Control + protein supplementation
  * Training in aquabike
  * Training in aquabike + protein supplementation
  * Bicycle training
  * Bicycle training + protein supplementation
  Interventions: Behavioral: Physical activity program : aquabike; Behavioral: Physical activity program : with protein supplementation
- Bicycle training (Experimental): Physical condition will be evaluated in obese patients before surgery and 1, 4, 6, 12, 18 and 24 months after surgery.
  Between 1 and 4 months after surgery, participants will be assigned to one of the postoperative care groups:
  * Control
  * Control + protein supplementation
  * Training in aquabike
  * Training in aquabike + protein supplementation
  * Bicycle training
  * Bicycle training + protein supplementation
  Interventions: Behavioral: Physical activity program : bicycle; Behavioral: Physical activity program : without protein supplementation
- - Bicycle training + protein supplementation (Experimental): Physical condition will be evaluated in obese patients before surgery and 1, 4, 6, 12, 18 and 24 months after surgery.
  Between 1 and 4 months after surgery, participants will be assigned to one of the postoperative care groups:
  * Control
  * Control + protein supplementation
  * Training in aquabike
  * Training in aquabike + protein supplementation
  * Bicycle training
  * Bicycle training + protein supplementation
  Interventions: Behavioral: Physical activity program : bicycle; Behavioral: Physical activity program : with protein supplementation

INTERVENTIONS:
Behavioral: Physical activity program : aquabike — The aim of this project is to investigate in obese patients the changes induced by bariatric surgery on the various components of the physical condition and their postoperative evolution following an intervention combining a physical activity program (aquabike vs bicycle) with or without protein supplementation.
  Arms: - Training in aquabike + protein supplementation; Training in aquabike
Behavioral: Physical activity program : bicycle — The aim of this project is to investigate in obese patients the changes induced by bariatric surgery on the various components of the physical condition and their postoperative evolution following an intervention combining a physical activity program (aquabike vs bicycle) with or without protein supplementation.
  Arms: - Bicycle training + protein supplementation; Bicycle training
Behavioral: Physical activity program : with protein supplementation — The aim of this project is to investigate in obese patients the changes induced by bariatric surgery on the various components of the physical condition and their postoperative evolution following an intervention combining a physical activity program (aquabike vs bicycle) with or without protein supplementation
  Arms: - Bicycle training + protein supplementation; - Training in aquabike + protein supplementation; Control + protein supplementation
Behavioral: Physical activity program : without protein supplementation — The aim of this project is to investigate in obese patients the changes induced by bariatric surgery on the various components of the physical condition and their postoperative evolution following an intervention combining a physical activity program (aquabike vs bicycle) with or without protein supplementation
  Arms: Bicycle training; Control; Training in aquabike

SUMMARY:
The aim of this project is to investigate in obese patients the changes induced by bariatric surgery on the various components of the physical condition and their postoperative evolution following an intervention combining a physical activity program (aquabike vs bicycle) with or without protein supplementation.

DETAILED DESCRIPTION:
Physical condition will be evaluated in obese patients before surgery and 1, 4, 6, 12, 18 and 24 months after surgery.

Between 1 and 4 months after surgery, participants will be assigned to one of the postoperative care groups:

* Control
* Control + protein supplementation
* Training in aquabike
* Training in aquabike + protein supplementation
* Bicycle training
* Bicycle training + protein supplementation

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Age between 18 and 60 years
* Body mass index: BMI> 40 kg / m2
* Candidates for bariatric surgery

Exclusion Criteria:

* Subject under 18 or over 60 years of age
* Biological assessment considered abnormal by the investigator
* HIV serology or known positive HCV
* Pregnant or nursing women
* For women of childbearing age: beta-hCG positive dosage or absence of contraception deemed reliable (oral contraceptive, IUD, implant or hormonal patch)
* Medical or surgical history (judged by the investigator to be inconsistent with the study)
* Subject with cardiorespiratory and / or osteo-articular disorders limiting their ability to perform physical tests or training
* Subject with cardiovascular or neoplastic disease
* Subjects with an infection in the 3 months prior to inclusion
* Hypercorticism and uncontrolled dysthyroidism
* Patient with known neuro-muscular pathology: myopathy, myasthenia gravis, rhabdomyolysis, paraplegia, hemiplegia
* Patient with chronic or acute inflammatory disease the 3 months before inclusion
* CRP> 20 mg / l
* Person treated with or having stopped treatment for less than 3 months prior to inclusion by corticosteroids, immunosuppressant, anabolic agent, growth hormone
* Person with an unstable psychiatric condition
* Blood donation in the two months preceding the study
* High alcohol consumption (> 2 to 3 drinks per day depending on sex) or presence of drug addiction
* Significant smoking (> 5 cigarettes / day or equivalent in cigars or pipe tobacco)
* Intense sports activity (> 5 hours / week)
* Subjects excluded from another study or having received more than 4500 € in the year following their participation in clinical studies

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-10-23 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Distance traveled at the 6-minute walking test (TM6) | at 4 months post-surgery

SECONDARY OUTCOMES:
Body composition | at 4 months post-surgery
resting metabolic rate | at 4 months post-surgery
VO2 max | at 4 months post-surgery
food consumption | at 4 months post-surgery
physical activity level | at 4 months post-surgery
muscle maximal strength evaluated by an isokinetic dynamometer | at 4 months post-surgery
evaluation of the equilibrium of the body on a stabilometric platform | at 4 months post-surgery
muscle typology | at 4 months post-surgery
muscle oxidative capacity | at 4 months post-surgery
muscle fat infiltration | at 4 months post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yves BOIRIE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France